CLINICAL TRIAL: NCT01382498
Title: Effect of Doxium on High Sensitivity CRP and Endothelin-1 Serum Levels in Patients With Diabetic Retinopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tabriz University (Other)
Responsible Party: Tabriz Medical University Biotechnology research center, Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 88-8
Record Dates: First submitted 2010-05-21; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-04

CONDITIONS: Diabetic Retinopathy
Keywords: Endothelin-1 high sensitivity CRP
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablets will be administered to the patients in Placebo arms daily for three months.
  Interventions: Drug: Placebo drug
- Calcium dobesilate (Experimental): Calcium dobesilate as 500 mg tablets will be administered once to the patients daily.
  Interventions: Drug: Calcium dobesilate (Doxium)

INTERVENTIONS:
Drug: Calcium dobesilate (Doxium) — 500 mg, Tablet, Daily, 3 months
  Arms: Calcium dobesilate
Drug: Placebo drug — Similar to the that of the Experimental arm, Daily, Three months
  Arms: Placebo

SUMMARY:
Diabetic retinopathy (DR) is a highly specific vascular complication of type 1 and type 2 diabetes mellitus. Calcium dobesilate(CD) or Doxium has been tested in the treatment of diabetic retinopathy showing a slowdown of the progression of the disease after long-term oral treatment,as a potent antioxidant. Endothelin-1 (ET-1) Besides being a very potent vasoconstrictor,acts as a mitogen on the vascular smooth muscle and play the main role in the failure of autoregulation that it is an important and often early feature of diabetic retinopathy.several studies have been confirmed that inflammation besides oxidative stress are the main mechanisms,in the pathogenesis of DR and hsCRP can play a sensitive role in detecting inflammation in these patients. The aim of this study was to determine the effects of CD on decreasing ET-1 and hsCRP serum levels in patients with diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* BS 120-200 mg/dl
* Age 40-70
* Severe NPDR(non proliferative diabetic retinopathy) or PDR(proliferative diabetic retinopathy)
* type II diabetes
* no history of doxium consumption

Exclusion Criteria:

* Allergy to doxium
* incidence of active hepatic disease or rising of hepatic enzymes during the intervention

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
high sensitivity CRP and Endothelin-1 serum levels | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Tabriz University of Medical Sciences, Tabriz, Eastern Azerbayjan, Iran